CLINICAL TRIAL: NCT05718271
Title: The Effects of Verbal Instructions on Fear Extinction and Extinction Retrieval in Patients With Anxiety Disorders and Healthy Controls
Brief Title: Effects of Verbal Instructions on Fear Extinction and Extinction Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Annalisa Lipp, M. Sc., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 673
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Anxiety Disorder
Keywords: anxiety disorders; fear extinction; fear conditioning; instructions; contingencies
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Explicit instructions before + after extinction (Experimental)
  Interventions: Other: Explicit instructions before extinction; Other: Explicit instructions after extinction
- Explicit instructions before extinction (Experimental)
  Interventions: Other: Explicit instructions before extinction
- Explicit instructions after extinction (Experimental)
  Interventions: Other: Explicit instructions after extinction
- No explicit instructions (No Intervention)

INTERVENTIONS:
Other: Explicit instructions before extinction — "Shocks will no longer be administered during the next phase."
  Arms: Explicit instructions before + after extinction; Explicit instructions before extinction
Other: Explicit instructions after extinction — "Tomorrow no shocks will be administered."
  Arms: Explicit instructions after extinction; Explicit instructions before + after extinction

SUMMARY:
The goal of this study is to examine if verbal instructions can improve fear extinction learning and extinction retrieval in patients with anxiety disorders (AD) and healthy controls.

DETAILED DESCRIPTION:
Patients with anxiety disorders (AD) and highly anxious individuals show accelerated fear conditioning and diminished fear extinction learning (Duits et al., 2015). The aim of the current study is to investigate how verbal instructions impact fear extinction learning and extinction retrieval in AD patients and healthy controls. Using a 3-day fear conditioning paradigm, fear acquisition will take place on the first, extinction training on the second, and extinction retrieval and reinstatement on the third day (i.e., all phases are on consecutive days). Part of the participants will receive explicit instructions such that the unconditioned stimulus (UCS) won't be presented anymore, either before and/or after extinction training. Participants will be randomly assigned to four conditions: (1) no explicit instructions at all, (2) explicit instructions before extinction, (3) explicit instructions after extinction or (4) explicit instructions before and after extinction.

ELIGIBILITY:
Inclusion Criteria:

* For the patient group: DSM-5 anxiety disorder diagnosis via a structured clinical interview for diagnosing mental disorders (DIPS)
* For the healthy controls: no psychological disorder according to the Mini-DIPS

Exclusion Criteria:

* smoking
* alcohol abuse
* drug consumption
* current and chronic physical and neurological diseases
* for the patient group: anxiety not the primary diagnosis, psychological comorbidities e.g. schizophrenia, bipolar disorder, mental retardation, acute drug or alcohol addiction, personality disorder, currently in psychotherapy
* for the healthy controls: a diagnosis of psychological disorder at any point in life, ever been in psychotherapy, current and/or regular intake of medicine (incl. psychopharmaceutic medicine), current or past cognitive or neurological disorder
* for women: pregnancy, nursing period
* previous experience with fear conditioning paradigm

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Fear extinction learning | Experimental Day 2
  The difference between the reinforced conditioned stimulus (CS+) and non-reinforced conditioned stimulus (CS-) will be measured on 3 different levels: skin conductance responses (SCRs), CS valence ratings ("How pleasant do you feel when you see this picture?"), and UCS expectancy ratings ("Do you think that this picture is paired with an electrical stimulation?").
Extinction retrieval | Experimental Day 3
  The difference between the reinforced conditioned stimulus (CS+) and non-reinforced conditioned stimulus (CS-) will be measured on 3 different levels: skin conductance responses (SCRs), CS valence ratings ("How pleasant do you feel when you see this picture?"), and UCS expectancy ratings ("Do you think that this picture is paired with an electrical stimulation?").

SECONDARY OUTCOMES:
Fear acquisition | Experimental Day 1
  The difference between the reinforced conditioned stimulus (CS+) and non-reinforced conditioned stimulus (CS-) will be measured on 3 different levels: skin conductance responses (SCRs), CS valence ratings ("How pleasant do you feel when you see this picture?"), and UCS expectancy ratings ("Do you think that this picture is paired with an electrical stimulation?").
Contingency awareness | Experimental Day 1
  After fear acquisition, it will be checked if participants can correctly determine which CS had been paired with the UCS.

OTHER OUTCOMES:
Score on Intolerance of Uncertainty Scale | Experimental Day 1
  The Intolerance of Uncertainty Scale measures a person's degree of vigilance, burden and disturbed action ability when experiencing uncertain situations. The items are scored on a 5-point scale from 1 = "not at all characteristic of me' to 5 = "entirely characteristic of me" and higher IU scale scores are related to higher intolerance of uncertainty. High IU supposedly plays an important role in maintaining fear and anxiety and is related to poorer fear extinction.
Score on General Self-efficacy (GSE) Scale | Experimental Day 1
  The GSE Scale contains ten items and measures how confident the person feels to overcome difficult situations based on their self-assessed competence. The GSE items are scored on a four-point scale with 1 = not at all true, 2 = hardly true, 3 = moderately true and 4 = exactly true. The total score is determined by summing up all item scores, which results in a score between 10 and 40, where the higher scores represent higher GSE.
Trait Anxiety score on State-Trait-Anxiety Inventory | Experimental Day 1
  Trait anxiety will be measured with 20 items of the State-Trait Anxiety Inventory. The items are measured on a four-point scale ranging from 1 = hardly ever to 4 = always. The total score of trait anxiety is calculated by summing up the scores (ranging from 20 to 80), whereby higher scores are indicative of higher trait anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zlomuzica, PhD, Principal Investigator — Ruhr University Bochum; Marcella L Woud, PhD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Ruhr University Bochum, Bochum, Germany

IPD SHARING:
Plan to Share IPD: Yes
This study is carried out within the framework of the German Research Foundation (DFG) funded Collaborative Research Center (SFB) 1280 "Extinction learning". Within the framework of the SFB, almost 20 research groups from Bochum, Essen and Dortmund are working together. Part of the collected data is evaluated jointly. For this purpose, part of the data (e.g. skin conductance, questionnaires) and general information about the person (e.g. gender, age, schooling) are passed on in a pseudonymized form to a central project. Pseudonymized means that the participant's name and date of birth will be replaced by a code and the assignment to the person is only available for employees of this study, but not for employees of the central project.

REFERENCES:
- [Background] Duits P, Cath DC, Lissek S, Hox JJ, Hamm AO, Engelhard IM, van den Hout MA, Baas JM. Updated meta-analysis of classical fear conditioning in the anxiety disorders. Depress Anxiety. 2015 Apr;32(4):239-53. doi: 10.1002/da.22353. Epub 2015 Feb 20. PMID 25703487